CLINICAL TRIAL: NCT06028178
Title: Clinical Evaluation of Droplet Digital Polymerase Chain Reaction in Combination With Transcriptome Analysis in Early Warning of Sepsis in the Emergency Department: A Multicenter Prospective Observational Study
Brief Title: Droplet Digital PCR Combines With Transcriptome Analysis in Early Warning of Sepsis in the Emergency Department
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai East Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: emergency medicine 20230824
Record Dates: First submitted 2023-08-17; First posted 2023-09-08 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2023-09

CONDITIONS: Sepsis; Emergent Infections, Treatment
Keywords: Droplet digital PCR; Transcriptomic molecular target assay
MeSH Terms: conditions — Sepsis; Breakthrough Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental group: The experimental group will recruit 300 participants undergoing blood culture, droplet digital PCR and transcriptome analysis.
  Interventions: Diagnostic Test: Droplet digital PCR
- Control group: The control group will recruit 60 participants undergoing blood culture only.

INTERVENTIONS:
Diagnostic Test: Droplet digital PCR — Droplet digital PCR has potential in resolving polymicrobial infection because it simultaneously achieves unprecedented high sensitivity , high specificity, and absolute quantification without the need for a standard curve.
  Other Names: Transcriptomic analysis
  Groups: Experimental group

SUMMARY:
Rapid identification of pathogens and early warning of host response are key to improve the prognosis of sepsis. Establishing a comprehensive identification system based on pathogen identification and host immune status is an effective way to achieve early warning stratification of patients with infections in the emergency department. This prospective multicenter clinical study will combine droplet digital PCR (ddPCR) and transcriptomic molecular target assay for validation in patients with suspected sepsis in the emergency department. The purpose is to (1) compare the efficacy of ddPCR with blood culture for early diagnosis and prognosis; (2) assess the diagnostic value of transcriptomic molecular targets based on 29 messenger RNA for the presence or absence of infection as well as infectious agents, and to evaluate their efficacy for prognosis; and (3) assess the diagnostic and therapeutic monitoring value of ddPCR combined with transcriptome analysis methods.

DETAILED DESCRIPTION:
Rapid identification of pathogens and early warning of host response are key to improve the prognosis of sepsis. Establishing a comprehensive identification system based on pathogen identification and host immune status is an effective way to achieve early warning stratification of patients with infections in the emergency department. Therefore, based on our preliminary single-center study, this prospective multicenter clinical study will combine droplet digital PCR (ddPCR) and transcriptomic molecular target assay for validation in patients with suspected sepsis in the emergency department. The purpose is to (1) compare the efficacy of ddPCR with blood culture for early diagnosis and prognosis; (2) assess the diagnostic value of transcriptomic molecular targets based on 29 messenger RNA for the presence or absence of infection as well as infectious agents, and to evaluate their efficacy for prognosis; and (3) assess the diagnostic and therapeutic monitoring value of ddPCR combined with transcriptome analysis methods. In a word, this study will be undertaken to assess the diagnostic and therapeutic monitoring value of early warning models for sepsis in emergency department and to promote them to improve the identification ability of emergency infections.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years, regardless of sex
* MSS≥2 score
* written informed consent obtained

Exclusion Criteria:

* Age < 18 years, regardless of sex
* Patient's ICU length of stay <24 hours
* Malignant tumor, HIV patients or any terminal-stage disease
* Known pregnancy or lactation
* Participation in other clinical trials
* Inadequate clinical information or missing experimental data
* No signed informed consent obtained

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective inclusion of patients with suspected sepsis with MSS ≥ 2 in the emergency department of Shanghai East Hospital, Shanghai Pudong New District Zhoupu Hospital, Shanghai Pudong New District Gongli Hospital, Shanghai Pudong Hospital and Shanghai Punan Hospital Hospital, Shanghai Pudong Hospital, Shanghai Pudong New Area Hospital and Shanghai Pudong New Area Punan Hospital. The patients will be randomized by stratified grouping and assigned to two parallel groups in the ratio of 5:1.
Sampling Method: Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic efficiency of ddPCR combined with transcriptomic analysis in suspected sepsis | 7days
  Diagnostic efficiency of ddPCR combined with transcriptomic analysis for suspected sepsis in the emergency medicine
Prognostic value of ddPCR combined with transcriptomic analysis in suspected sepsis | 28 days
  Prognostic value of ddPCR combined with transcriptomic analysis for suspected sepsis in the emergency medicine

SECONDARY OUTCOMES:
7-day all-cause mortality rate | 7 days
  Evaluation of combined examination by ddPCR and transcriptomic analysis for the evaluation of the prognosis of the sepsis.
28-day all-cause mortality rate | 28 days
  Evaluation of combined examination by ddPCR and transcriptomic analysis for the evaluation of the prognosis of the sepsis.
90-day all-cause mortality rate | 90 days
  Evaluation of combined examination by ddPCR and transcriptomic analysis for the evaluation of the prognosis of the sepsis.
Antimicrobial Resistance and antibiotic application | 7 days
  Evaluation of combined examination by ddPCR and transcriptomic analysis for the the value of guiding clinical drug therapy.

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 3 years